CLINICAL TRIAL: NCT03112590
Title: A Phase I-II Study of Interferon-gamma Plus Weekly Paclitaxel, Trastuzumab and Pertuzumab in Patients With HER-2 Positive Breast Cancer
Brief Title: Phase I-II Study of Interferon-gamma in Patients With HER-2 Positive Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Horizon Pharma Ireland, Ltd., Dublin Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18936
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Results first posted 2022-06-08 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Breast Cancer, Male; Breast Cancer Female; HER2-positive Breast Cancer
Keywords: Histologically confirmed HER2 positive breast cancer; Unresectable breast cancer; Locally advanced breast cancer; Metastatic breast cancer; Clinical stage 2-3 early stage breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Interferon-gamma; interferon gamma-1b; Paclitaxel; Albumin-Bound Paclitaxel; Trastuzumab; pertuzumab; Antibodies, Monoclonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination Therapy (Experimental): Phase 1: Participants with HER-2 positive metastatic breast cancer enrolled in groups of 3-6 or more; each group participant to be given the same dose and schedule of Interferon-gamma plus paclitaxel, trastuzumab, and pertuzumab. If group participants do not have bad side effects, the next group will be given a higher dose of Interferon-gamma. This will continue until the highest safe dose of Interferon-gamma is found. Once highest safe dose of Interferon-gamma is found, participants may be enrolled in Phase II.
  Phase 2: Approximately 31 participants with Stage 2-3 HER2 positive early stage breast cancer enrolled to receive therapy with Interferon-gamma plus paclitaxel, trastuzumab, and pertuzumab. Interferon-gamma given at dose found in the Phase 1.
  Phase 2: Post therapy surgery.
  Interventions: Biological: Interferon-gamma (IFN-γ); Drug: Paclitaxel; Drug: Trastuzumab; Other: Pertuzumab; Procedure: Post Therapy Surgery

INTERVENTIONS:
Biological: Interferon-gamma (IFN-γ) — Phase 1: IFN-γ 50 or 75 mcg/m^2 SQ x 3 days/week for 12 weeks. Phase 2: IFN-γ at Recommended Phase II Dose (RP2D) subcutaneously (SQ) x 3 days/week, for 12 weeks.
  Other Names: Actimmune®; signaling proteins
Drug: Paclitaxel — Phase 1 and Phase 2: Paclitaxel 80 mg/m^2/week, for 12 weeks.
  Other Names: Abraxane®
Drug: Trastuzumab — Phase 1 and Phase 2: Trastuzumab 8 mg/kg intravenous (IV) loading dose on cycle 1/day 1 (C1D1), followed by 6 mg/kg on subsequent cycles every 3 weeks, for 12 weeks.
  Other Names: Herceptin®
Other: Pertuzumab — Phase 1 and Phase 2: Pertuzumab 840 mg IV loading dose on C1D1, followed by 420 mg on subsequent cycles every 3 weeks, for 12 weeks.
  Other Names: PERJETA®; monoclonal antibody
Procedure: Post Therapy Surgery — Phase 2: Participants will be assessed for surgery following the fourth cycle of study therapy (or earlier if study treatment is cancelled due to unmanageable side effects).

SUMMARY:
This purpose of this study is to evaluate the safety and to find the optimal dose in participants with human epidermal growth factor receptor 2 (HER2) positive breast cancer who are given the combination of Interferon-gamma with paclitaxel, trastuzumab and pertuzumab. This study will also look at other effects of Interferon-gamma with paclitaxel, trastuzumab and pertuzumab, including its effect on this type of cancer.

Interferon-gamma is a biologically manufactured protein that is similar to a protein the body makes naturally. In the body, interferon gamma is produced by immune cells and helps to prevent serious infections.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histologically confirmed HER2 positive breast cancer (by ImmunoHistoChemistry (IHC) 3+ or fluorescence in situ hybridization (FISH) ratio ≥ 2.0). Phase 1: unresectable locally advanced or metastatic breast cancer. Phase 2: clinical stage 1-3 early stage breast cancer with primary tumor is at least 1cm measured by clinical exam or by radiologic breast imaging tests.
* Prior Therapy - Phase 1: Must be candidates to receive paclitaxel chemotherapy in combination with trastuzumab and pertuzumab. Phase 2: No prior chemotherapy, radiation, or definitive therapeutic surgery (e.g., mastectomy, lumpectomy or axillary dissection) for this malignancy. Patients who have had a prior sentinel lymph node biopsy for this malignancy are eligible. Patients who received equal to or less than 1 cycle of therapy (up to 4 weeks) will be allowed to enroll in this trial.
* Patients who received tamoxifen or another selective estrogen receptor modulator (SERM) for the prevention or treatment of breast cancer or for other indications (e.g., osteoporosis, prior ductal carcinoma in situ (DCIS)), or who receive aromatase inhibitors for prevention or treatment of breast cancer, are eligible. Patients who are hormone-receptor positive and who have received other hormonal agents for the treatment of breast cancer (e.g., Fulvestrant®) are also eligible. Tamoxifen therapy or other hormonal agents should be discontinued at least 1 week before the patient is started on study therapy.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Must have normal organ and marrow function within 2 weeks of registration (except where specified otherwise).
* Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Receiving any other investigational agents during protocol therapy, or up to 14 days or 5 half-lives (whichever is longer) prior to beginning protocol therapy. There should be a least a 1-week interval between last dose of endocrine therapy and protocol therapy.
* Have had chemotherapy or radiation therapy within 2 weeks prior to beginning protocol therapy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, congenital prolonged QT syndrome, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Current use of corticosteroid therapy > 5 mg/day of prednisone or equivalent doses of other corticosteroids (topical, intranasal, and inhaled corticosteroids in standard doses and physiologic replacement for participants with adrenal insufficiency are allowed).
* Known active or symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis. Asymptomatic, treated, and/or stable brain metastases, as measured by subsequent radiologic evaluations at least two months apart, are permitted.
* Pregnant or breast feeding.
* Known HIV-positive.
* Known current or a history of hepatitis B or C virus, including chronic and dormant states, unless disease has been treated and confirmed cleared.
* Major surgery within 4 weeks of initiation of study drug.
* Second invasive malignancy requiring active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2023-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: (Hyo) Heather S. Han, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Gautam N, Elleson KM, Ramamoorthi G, Czerniecki BJ. Current State of Cell Therapies for Breast Cancer. Cancer J. 2022 Jul-Aug 01;28(4):301-309. doi: 10.1097/PPO.0000000000000607. PMID 35880940
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/
- See also: Residual Cancer Burden (RCB) — http://www3.mdanderson.org/app/medcalc/index.cfm?pagename=jsconvert3

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Level 1: Interferon-gamma (IFN-γ): Phase 1: IFN-γ 50 mcg/m^2 SQ x 3 days/week for 12 weeks.
  Paclitaxel: Phase 1 and Phase 2: Paclitaxel 80 mg/m^2/week, for 12 weeks.
  Trastuzumab: Phase 1 and Phase 2: Trastuzumab 8 mg/kg intravenous (IV) loading dose on cycle 1/day 1 (C1D1), followed by 6 mg/kg on subsequent cycles every 3 weeks, for 12 weeks.
  Pertuzumab: Phase 1 and Phase 2: Pertuzumab 840 mg IV loading dose on C1D1, followed by 420 mg on subsequent cycles every 3 weeks, for 12 weeks.
- Phase 1 Level 2: Interferon-gamma (IFN-γ): Phase 1: IFN-γ 75 mcg/m^2 SQ x 3 days/week for 12 weeks.
  Paclitaxel: Phase 1 and Phase 2: Paclitaxel 80 mg/m^2/week, for 12 weeks.
  Trastuzumab: Phase 1 and Phase 2: Trastuzumab 8 mg/kg intravenous (IV) loading dose on cycle 1/day 1 (C1D1), followed by 6 mg/kg on subsequent cycles every 3 weeks, for 12 weeks.
  Pertuzumab: Phase 1 and Phase 2: Pertuzumab 840 mg IV loading dose on C1D1, followed by 420 mg on subsequent cycles every 3 weeks, for 12 weeks.
- Phase 2: Interferon-gamma (IFN-γ): Phase 2: IFN-γ 75 mcg/m^2 SQ x 3 days/week for 12 weeks.
  Paclitaxel: Phase 1 and Phase 2: Paclitaxel 80 mg/m^2/week, for 12 weeks.
  Trastuzumab: Phase 1 and Phase 2: Trastuzumab 8 mg/kg intravenous (IV) loading dose on cycle 1/day 1 (C1D1), followed by 6 mg/kg on subsequent cycles every 3 weeks, for 12 weeks.
  Pertuzumab: Phase 1 and Phase 2: Pertuzumab 840 mg IV loading dose on C1D1, followed by 420 mg on subsequent cycles every 3 weeks, for 12 weeks.
Period: Overall Study
Arm/Group | Phase 1 Level 1 | Phase 1 Level 2 | Phase 2
Started | 3 | 6 | 42
Completed | 3 | 5 | 42
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Level 1 | Phase 1 Level 2 | Phase 2 | Total
Number analyzed (Participants) | 3 | 6 | 42 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 28 | 37
  >=65 years | 0 | 0 | 14 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 42 | 51
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 5 | 5
  Not Hispanic or Latino | 3 | 6 | 37 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 3 | 3 | 37 | 43
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 42 | 51

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Recommended Phase 2 Dose (RP2D)
Description: The dose limiting toxicity (DLT) evaluation period for dose escalation will be during the first three weeks. The maximum tolerated dose (MTD) dose level is defined as the highest dose level with ≤1 out of 6 participants experiencing a DLT. If the first dose level experience two or more DLTs, then dose de-escalation will occur. DLT during cycle one (C1) is defined as follows: Non-hematologic or hematologic toxicities that are ≥ grade 3 in severity and probably or definitely related to study therapy which leads to chemotherapy treatment delays > 14 days are considered DLT. The MTD will become the RP2D.
Time Frame: 12 weeks
Measure: Number; unit: mcg/m^2
Groups:
- Combination Therapy: Interferon-gamma (IFN-γ): Phase 1: IFN-γ 50 or 75 mcg/m^2 SQ x 3 days/week for 12 weeks.
  Phase 2: IFN-γ at Recommended Phase II Dose (RP2D) subcutaneously (SQ) x 3 days/week, for 12 weeks.
  Paclitaxel: Phase 1 and Phase 2: Paclitaxel 80 mg/m^2/week, for 12 weeks.
  Trastuzumab: Phase 1 and Phase 2: Trastuzumab 8 mg/kg intravenous (IV) loading dose on cycle 1/day 1 (C1D1), followed by 6 mg/kg on subsequent cycles every 3 weeks, for 12 weeks.
  Pertuzumab: Phase 1 and Phase 2: Pertuzumab 840 mg IV loading dose on C1D1, followed by 420 mg on subsequent cycles every 3 weeks, for 12 weeks.
Arm/Group | Combination Therapy
Number analyzed (Participants) | 9
mcg/m^2 | 75

2. Primary Outcome: Phase 2: Pathologic Complete Response Rate (pCR)
Description: Pathologic complete response in the breast at definitive surgery after completion of protocol therapy. The pathologic response to treatment will be assessed by an institutional pathologist at Moffitt Cancer Center. The pathologist will evaluate response by the "Residual Cancer Burden"(RCB) for each participant as described in the online calculator (see RCB link in the More Information section). pCR is defined as no residual invasive carcinoma in the breast and lymph notes at definitive surgery following neoadjuvant therapy
Time Frame: After post therapy surgery - Therapy: approximately 12 weeks per participant
Population: Evaluable participants
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 23
percentage of participants | 52

3. Secondary Outcome: Phase 2: Clinical Response
Description: Complete Response (CR) and Partial Response (PR) based upon tumor measurements obtained on physical examination at baseline, after completion of 4 cycles of study therapy. Factors that will be evaluated include: Breast mass(es) - size (longest dimension); Axillary lymph node(s) - size (longest dimension); Skin edema of the breast - present worse, present unchanged, present improved, or absent; Skin erythema of the breast - present worse, present unchanged, present improved, or absent.
Time Frame: 12 weeks
Population: Evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2
Number analyzed (Participants) | 39
Participants
  Complete Response | 25
  Partial Response | 11
  Stable Disease | 2
  Progressive Disease | 1

4. Secondary Outcome: Phase 2: Progression Free Survival (PFS)/Number of Participants Who Progressed
Description: Progression will be evaluated in this study using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria, version 1.1.
  PFS is defined as the time from study therapy to the first occurrence of ipsilateral invasive breast tumor recurrence, ipsilateral locoregional invasive breast cancer recurrence, contralateral invasive breast cancer, distant recurrence, or death from any cause. This is reported as number of participants who progressed.
Time Frame: Up to 2 years
Population: Evaluable participants
Measure: Number; unit: participants
Arm/Group | Phase 2
Number analyzed (Participants) | 39
participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from date of on study to 30 days after last dose of study treatment, up to 4 months.
Arm/Group | Phase 1 Level 1 | Phase 1 Level 2 | Phase 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/6 | 2/42
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 4/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Level 1 (N=3) | Phase 1 Level 2 (N=6) | Phase 2 (N=42)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Level 1 (N=3) | Phase 1 Level 2 (N=6) | Phase 2 (N=42)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 1 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 2 (2) | 1 (1)
Fever (General disorders) | 1 (1) | 3 (4) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal disorders -Other (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — worsening
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 3 (3) | 2 (4)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — deep cut
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Movements involuntary (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Restless legs
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (7)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — Skin lesions
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 2 (4) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — rhinorrhea
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT03112590/Prot_SAP_000.pdf